CLINICAL TRIAL: NCT06908226
Title: A Phase 3, Open-Label Study to Investigate the Long-Term Safety and Efficacy of LP352 in the Treatment of Seizures in Children and Adults With Developmental and Epileptic Encephalopathy
Brief Title: A Study to Investigate LP352 in Children and Adults With Developmental and Epileptic Encephalopathy (DEE)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Longboard Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP352-303; 2024-514974-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-06; First posted 2025-04-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Developmental and Epileptic Encephalopathy
Keywords: Developmental and Epileptic Encephalopathy; LP352; Bexicaserin; Seizures; DEEp OLE; Antiseizure medications; Epilepsy; Neurodevelopmental disorders; Dravet syndrome; Lennox-gastaut syndrome
MeSH Terms: conditions — Seizures; Epilepsy; Neurodevelopmental Disorders; Epilepsies, Myoclonic; Lennox Gastaut Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LP352 (Experimental): Participants will be titrated up to highest tolerated dose of LP352 during the Titration period (Visit 1 - Visit 3), followed by maintenance period (Visit 4 - Visit 14) and then taper/down titration period (Visit 15 - Visit 17).
  Interventions: Drug: LP352

INTERVENTIONS:
Drug: LP352 — LP352 will be administered orally or through G-tube/ percutaneous endoscopic gastrostomy (PEG) tube.
  Other Names: Bexicaserin

SUMMARY:
This (DEEp OLE Study) is a multicentre, open-label study to investigate the long-term safety, efficacy, tolerability, and pharmacokinetics (PK) of LP352 in the treatment of seizures in children and adults with DEE who completed Study LP352-301 or LP352-302. The study consists of 3 main phases: Screening, Titration period and Maintenance period, followed by a Taper period and Follow-Up. The total duration of the study will be approximately 14 months.

ELIGIBILITY:
Inclusion Criteria:

* The participant has satisfactorily completed Study LP352-301 or LP352-302 Visit 8, and who, in the opinion of the investigator, may benefit from continued LP352 administration.
* Diagnosis of DEE that includes Dravet Syndrome (DS), Lennox-Gastaut Syndrome (LGS), or DEE Other (as defined and evaluated in Study LP352-301 or LP352-302).
* Participant has a body weight of ≥10 kg.
* G-tubes/PEG tubes (if applicable) should be in stable and good working condition. Nasogastric tubes are not allowed except for short-term management.
* Has at least one reliable and consistent parent, legal guardian, or caregiver during the study.
* The participant must be willing and able to provide written informed consent; in instances where the participant is unable to provide consent, an appropriate LAR must provide informed consent and the participant will need to assent (as per local regulations) before participation in the study. If the participant cannot provide consent or assent (ie, due to developmental status), the investigator should document why it was not obtained.
* The participant and/or authorized representative is willing to provide written consent or assent to allow the investigator and the investigator's staff to consult with the participant's medical caregivers and the medical monitor during Screening and during participation in the study.
* All participants of childbearing potential must have a negative urine or serum pregnancy (human chorionic gonadotropin) test at Visit 8 from Study LP352-301 or LP352-302 and agrees to routinely use an acceptable effective method of contraception from the time of signing informed consent up to 48 hours after the last dose of study drug.
* Participant and/or participant's caregiver(s) agree to not post any participant's personal medical data related to the study or information related to the study on any website or social media site until the study has been completed.
* The participant, parent, or caregiver is willing and able (in the judgment of the investigator) to comply with completion of the diaries throughout the study.

Exclusion Criteria:

* The participant is receiving exclusionary medications.
* Considered at risk of suicidal behavior based on the C-SSRS at Visit 8 of LP352-301 or LP352-302. If the participant is unable to complete the C-SSRS due to developmental status, the participant's LAR may not complete the C-SSRS. In these cases, the investigator may use clinical judgment to assess both the participant's status regarding suicidality and the ability to complete the scale, both of which must then be documented in the source document.
* Has a PHQ-9 score of >9 or a positive response to Question 9 at Visit 8 of LP352-301 or LP352-302. If the participant is unable to complete the PHQ-9, the participant's LAR may not complete the PHQ-9. In these cases, the investigator may use clinical judgment to assess both the participant's status and ability to complete the scale, both of which must then be documented in the source document.
* Ongoing AE from LP352-301 or LP352-302 of severe depression, anorexia nervosa, or bulimia per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition.
* Has an abnormal and clinically significant 12-lead ECG at Visit 8 in LP352-301 or LP352-302 in the opinion of the investigator, for example, second- or third-degree heart block or a QTc of >450 msec for adult males, >470 msec for adult females, or >440 msec for pediatric participants.
* Ongoing AE in LP352-301 or LP352-302 of alcohol, opioid, or other drug use disorder, as per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition.
* Current use of any cannabis product or cannabidiol that is not in oral solution/capsule/tablet form, not obtained from a government-approved dispensary, or containing ≥50% THC. Cannabis product or cannabidiol should be used primarily to treat seizures and dose should not be adjusted for the duration of the study. Cannabis product or cannabidiol will count as a concurrent ASM.
* Has a positive result on the urine drug screen at Visit 8 of LP352-301 or LP352-302, except for positive results related to prescribed controlled medications (eg, benzodiazepine) or Epidiolex®/government-approved cannabis product/cannabidiol used to treat seizures (eg, tetrahydrocannabinol).
* Unstable, clinically significant neurologic (other than the disease being studied, eg, recurrent strokes), psychiatric, cardiovascular (eg, pulmonary arterial hypertension, cardiac valvulopathy, orthostatic hypotension/tachycardia) pulmonary, hepatic (severe hepatic impairment), renal (severe renal impairment), metabolic, gastrointestinal, urologic, immunologic, hematopoietic, or endocrine disease or other abnormality at Visit 8 of LP352-301 or LP352-302 which may impact the ability of the participant to participate or potentially confound the study results.
* Is pregnant, breast-feeding, or intending to become pregnant during or within 48 hours after the last dose of study drug; or intending to donate ova during such time period.
* Has a known hypersensitivity to any component of LP352 formulation or any history of serious drug-induced hypersensitivity, eg, toxic epidermal necrolysis or Drug Reaction with Eosinophilia and Systemic Symptoms.
* Unwilling to abstain from donation of blood during and within 2 weeks after the study.
* Is unable or unwilling to comply with any of the study requirements or timelines.

Ages: 2 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2027-11-11 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting Treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) and AEs leading to discontinuation | Up to 61 Weeks
  An AE is defined as any untoward medical occurrence in a participant enrolled into this study, regardless of its causal relationship to the study drug. A treatment-emergent AE is defined as any event that is not present before exposure to study drug or any event or condition that is already present that worsens in either intensity or frequency after exposure to study drug. An SAE is defined as any event that: Results in death; Is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization. "Inpatient hospitalization" includes admission to an emergency room for observation and/or treatment that would have been insufficient in an outpatient setting; results in persistent or significant disability/incapacity; Is a congenital anomaly/birth defect or is an important medical event. An adverse event of special interest (AESI) is an AE or SAE is defined as an AE or SAE of scientific or medical concern specific to the sponsor's product or program.
Number of Participants With Clinically Significant Changes in Chemistry parameters | Up to 61 Weeks
Number of Participants With Clinically Significant Changes in Hematology parameters | Up to 61 Weeks
Number of Participants With Clinically Significant Changes in Urinalysis | Up to 61 Weeks
Number of participants with clinically significant changes in vital signs | Up to 61 Weeks
Number of participants with clinically significant changes in physical examinations | Up to 61 Weeks
Number of participants with clinically significant changes in growth parameters | Up to 61 Weeks
Number of participants with clinically significant changes in electrocardiogram (ECG) parameters | Up to 61 Weeks
Number of participants with postive responses to Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 61 Weeks
  C-SSRS was developed by researchers at Columbia University as a tool to help systematically assess suicidal ideation and behavior. It is composed of questions addressing suicidal ideation and suicidal behavior, as well as self-injurious behavior without suicidal intent. The tool will be administered by a trained operator/interviewer (investigator or designee) via interview with the participant at the study time points. If the participant is unable to complete the C-SSRS due to developmental status, the participant's legally acceptable representative may not complete the C SSRS. In these cases, the investigator may use clinical judgment to assess both the participant's status regarding suicidality and ability to complete the scale, both of which must then be documented in the source document.
Number of participants with positive responses to Patient Health Questionnaire-9 (PHQ-9) and Question 9 | Up to 61 Weeks
  The PHQ-9 is a multipurpose instrument for Screening, diagnosing, monitoring, and measuring the severity of depression. The scale is an easy-to-use participant questionnaire that is a self-administered version of the Primary Care Evaluation of Mental Disorders diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 Diagnostic and Statistical Manual of Mental Disorders IV, Text Revision criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care. Participants with a depression score of greater than 9 (mild) on the PHQ-9 scale or a positive response to Question 9 should be excluded from the study. When there is a positive response to PHQ-9 Question 9 post randomization, the investigator should determine whether an AE has occurred.

SECONDARY OUTCOMES:
Frequency Percent Change in Countable Motor Seizures During Treatment Compared to Baseline | Baseline and up to 55 weeks
  The percent change from Baseline in countable motor seizure frequency during Treatment will be calculated as (countable motor seizure frequency during Treatment) - (countable motor seizure frequency during Baseline [Visit 1 of LP352-301 and LP352-302]) ÷ seizure frequency during Baseline [Visit 1 of LP352-301 and LP352-302]) × 100
Percentage of participants with ≥ 50% Reduction in countable motor seizures during Treatment compared to Baseline [Visit 1 of LP352-301 and LP352-302] | Baseline and up to 55 weeks
Frequency Percent Change in Countable Motor Seizures during Maintenance compared to Baseline [Visit 1 of LP352-301 and LP352-302] | Baseline and up to 55 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (9):
  - Arkansas Children's Hospital - PIN, Little Rock, Arkansas
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Research Institute of Orlando LLC, Orlando, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Institute of Neurology and Neurosurgery at Saint Barnabas, LLC, Livingston, New Jersey
  - Northeast Regional Epilepsy Group - Morristown - 310 Madison Ave, Morristown, New Jersey
  - The University of Texas Medical School at Houston, Houston, Texas
- Austin Hospital, Heidelberg, Victoria, Australia
- AP-HP - Hôpital universitaire Robert-Debré, Paris, France
- Children's Clinical University Hospital, Riga, Latvia
- Mother and Child Health Care Institute of Serbia Dr Vukan Cupic, Belgrade, Serbia
- Spain (3):
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vithas Madrid La Milagrosa, Madrid
  - Hospital Ruber Internacional (Grupo Quironsalud), Madrid

IPD SHARING:
Plan to Share IPD: Undecided